CLINICAL TRIAL: NCT05613296
Title: Real World Evaluation Among Italian Centers of the Activity and Safety of Fostamatinib in Consecutive Adult Patients With Immune Thrombocytopenia (ITP)
Brief Title: Real World Evaluation of the Activity and Safety of Fostamatinib in Consecutive Adult Patients With ITP
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ITP1122
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: ITP - Immune Thrombocytopenia; Chronic ITP; Refractory ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients being observed during the study duration.
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Patients with Chronic ITP, refractory to other treatment who received at least one dose of Fostamatinib outside clinical trials in Italy will be enrolled and observed for at least 6 months.

SUMMARY:
This is a retrospective and prospective multicenter observational study with the aim to evaluate the real-life use of Fostamatinib in adult patients with chronic ITP, refractory to other treatments.

DETAILED DESCRIPTION:
This is a retrospective and prospective multicenter observational study with the aim to evaluate the real-life use of Fostamatinib in adult patients with chronic ITP, refractory to other treatments.

All patients who received at least one dose of Fostamatinib between October 1st, 2021 and April 1st, 2023 outside interventional clinical trials in Italy in the participating centers will be invited to participate in the study. Every patient will be observed for at least 6 months until October 1st, 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic ITP who are refractory to other treatments and who received Fostamatinib according to standard clinical practice between October 1st, 2021 and April 1st, 2023
2. Age greater or equal to 18 years at the treatment start
3. Signed written informed consent document (if feasible) according to ICH/EU/GCP and national local laws

Exclusion Criteria:

1. Contraindications or hypersensitivity to Fostamatinib, its active substance or any of its excipients
2. Patients participating in an interventional clinical trial at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult ITP patients, refractory to other treatment, who received at least one dose of Fostamatinib between October 1st, 2021 and April 1st, 2023 outside interventional clinical trials in Italy in the participating Centers will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of ITP patients who receive Fostamatinib | 6 months
  effectiveness evaluation of fostamatinib

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Principal Investigator — Ematologia ASUGI Trieste
Locations (21):
- Italy (21):
  - AON SS. ANTONIO E BIAGIO E C. ARRIGO - SS emostasi e trombosi, Alessandria
  - SOD Clinica Ematologica AOU Ospedali Riuniti Umberto I GM Lancisi G Salesi, Ancona
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" Policlinico S. Orsola, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Unità di Onco-Ematologia - Azienda Ospedaliera Garibaldi, Catania
  - Ematologia A.O.U. Careggi, Florence
  - Milano Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia, Milan
  - Ematologia AOU Università degli Studi di Napoli "Federico II", Napoli
  - .C.D.U. Ematologia - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Aou Policlinico P. Giaccone Uo Ematologia, Palermo
  - Casa Di Cura La Maddalena S.P.A. - Dipartimento Oncologico Di Iii Livello - Uo Oncoematologia E Tmo, Palermo
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - S.C. di Ematologia, Arcispedale Santa Maria Nuova I.R.C.C.S., Reggio Emilia
  - Aou Policlinico Tor Vergata Uoc Trapianto Cellule Staminali, Roma
  - Fondazione P.U. Agostino Gemelli Irccs - Area Ematologica, Roma
  - Divisione di Ematologia "Città della Salute e della Scienza di Torino", Torino
  - Azienda Ospedaliera "Cardinale G. Panico", Ematologia e Centro Trapianti midollo osseo, Tricase
  - Clinica Ematologica-Azienda Sanitaria Universitaria Integrata di Trieste, Trieste
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - ULSS N.6 Ospedale S. Bortolo - Ematologia, Vicenza